CLINICAL TRIAL: NCT03934866
Title: The SUMMIT Study: Cancer Screening Study With or Without Low Dose Lung CT to Validate a Multi-cancer Early Detection Test
Brief Title: The SUMMIT Study: A Cancer Screening Study
Acronym: SUMMIT
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: GRAIL, Inc. (Industry); University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: UCL/17/0050
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken at each visit and sent to GRAIL to clinically validate a blood test for detecting multiple cancers at an early stage. An additional blood sample will be collected for (and stored by) UCL for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A (LDCT): 25,000 individuals who are at high-risk for lung cancer due to a significant smoking history.
  Participants will receive at least 1 LDCT scan at baseline.
  Interventions: Radiation: Low Dose CT scan

INTERVENTIONS:
Radiation: Low Dose CT scan — Low Dose chest CT scan conferring an equivalent radiation dose of less than 2 mSv to the average size patient. The study aims to keep most scans under 1 mSv (ultra-low dose), and all scans under 2 mSv.

SUMMARY:
The SUMMIT Study will enrol 13,000 participants in order to investigate how cancer screening can be improved and delivered. The SUMMIT Study has two main aims: the first is to clinically validate a blood test for detecting multiple cancers at an early stage. The second is to examine the feasibility of delivering a low-dose CT (LDCT) screening service for lung cancer to a high-risk population in North Central and East London.

DETAILED DESCRIPTION:
The SUMMIT Study is a prospective, observational, cohort study. Its aim is to clinically validate a blood test for the early detection of multiple types of cancer, and to deliver LDCT screening for lung cancer to an at-risk population.

SUMMIT plans to enrol 13,000 participants aged 55-77 years, from participating general practitioner (GP) practices in North Central and East London. The participants enrolled will be people who are at high-risk for lung cancer due to a significant smoking history based on validated risk scores.

Individuals with significant smoking histories will be offered a clinical Lung Health Check (LHC), which includes a brief respiratory consultation including questions about respiratory symptoms and medical history, smoking cessation advice and referral where required, and certain relevant clinical measurements (blood pressure, spirometry, height, and weight). Those persons who are eligible for participation based on specific validated risk scores may then be offered participation in the SUMMIT Study. Electronic informed consent will be obtained if they decide to take part. Consented participants will provide a blood sample, complete a confidential electronic questionnaire and have an LDCT scan at the same visit. Participants will be asked to return for two further annual visits, and some participants may return for additional scans if clinically indicated (nodule management).

If any LDCT result is suspicious for cancer, the participant will be referred to their local hospital (type 2 Site) via an urgent referral pathway to the relevant MDT. If a participant is diagnosed with lung cancer, that participant will no longer continue in the active/interventional part of the study but will be followed for clinical outcomes via the Type 2 site completion of eCRF and registry data. If the suspicious lesion is found to be benign, the participant can continue in the study.

There will be one randomisation round carried out during this study. All participants with a negative LDCT at the baseline visit who have not been diagnosed with lung cancer since that visit will return for an LHC at approximately 12 months. At the 12-month visit, this group will be randomised either to have an LDCT or no LDCT.

However, if an urgent referral was after the Y0 LDCT scan, the participant will not be included in the randomisation at Y1, and will receive LDCT at Y1 and Y2.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 55 to 77 years old at the time of GP data extraction, who meet either of the following criteria:

   1. USPSTF LDCT screening criteria: a history of at least 30 pack years of smoking and if a former smoker, have quit in the past 15 years; or
   2. PLCOm2012 6-year lung cancer risk of ≥1.3%
2. Capable of providing informed consent and willing to comply with all parts of the protocol

Exclusion Criteria:

Currently receiving treatment (e.g., chemotherapy, radiotherapy, watchful waiting) for an active cancer. If on adjuvant hormonal therapy can be included (e.g. for breast and prostate cancer).

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SUMMIT plans to enrol 13,000 participants, aged 55-77 years, from participating GP practices in north and east London who are at high-risk for lung cancer due to a significant smoking history.
Sampling Method: Non-Probability Sample
Enrollment: 13035 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the performance of the cell-free nucleic acid (cfNA) signals measured using high-intensity sequencing (ultra-deep and ultra-broad) for the detection of invasive cancer and identification of tissue of cancer origin using a GRAIL blood test. | 12 months
  Cancer incidence associated with screening test performance:
  * Sensitivity
  * False positive rate (1-specificity), specificity
  * Positive predictive value (PPV)
  * Negative predictive value (NPV)
To examine the performance of delivering a Low-Dose Computed Tomography (LDCT) screening service using established measures of performance and risk prediction of lung cancers and other incidental findings (see the performance indicators measured below). | 36 months
  Performance indicators that will be measured include the number of:
  * eligible participants who choose to have an LDCT.
  * characteristics of those who choose to have LDCT, e.g. age, sex, ethnicity, area-level deprivation score and smoking status.
  * people who have a baseline LDCT who attend at year 1 and also at year 2.
  * screen-detected cancers per 1000 screened
  * early stage screen-detected cancers per 1000 screened
  * late stage screen-detected cancers per 1000 screened
  * people referred for diagnostic investigations per 1000 screened
  * people who have a biopsy per 1000 screened
  * malignant and benign tumours detected
  * incidence per 1000 per year

CONTACTS AND LOCATIONS:
Locations (1):
- UCLH, London, United Kingdom

REFERENCES:
- [Derived] Mullin ML, Verghese P, Khaw CR, Creamer A, Bhamani A, Prendecki R, Dickson JL, Horst C, Tisi S, Hall H, Gyertson K, Arthur-Darkwa E, Farrelly L, McCabe J, Thakrar R, Nair A, Devaraj A, Navani N, Hackshaw A; SUMMIT consortium; Janes SM. Upstaging of screen-detected lung cancers during diagnostic assessment. Thorax. 2026 Feb 2:thorax-2025-224006. doi: 10.1136/thorax-2025-224006. Online ahead of print. PMID 41629156
- [Derived] Bhamani A, Creamer A, Verghese P, Prendecki R, Horst C, Tisi S, Hall H, Khaw CR, Mullin M, McCabe J, Gyertson K, Bowyer V, Arancon D, Eng J, Bojang F, Levermore C, Hacker AM, Arthur-Darkwa E, Farrelly L, Patel A, Lock S, Shaw A, Banka R, Bhowmik A, Ekeowa U, Mangera Z, Valerio C, Ricketts WM, Mohammed A, O'Shaughnessy T, Navani N, Quaife SL, Nair A, Devaraj A; SUMMIT consortium; Dickson JL, Hackshaw A, Janes SM. Low-dose CT for lung cancer screening in a high-risk population (SUMMIT): a prospective, longitudinal cohort study. Lancet Oncol. 2025 May;26(5):609-619. doi: 10.1016/S1470-2045(25)00082-8. Epub 2025 Mar 25. PMID 40154514
- [Derived] Tisi S, Creamer AW, Dickson J, Horst C, Quaife S, Hall H, Verghese P, Gyertson K, Bowyer V, Levermore C, Hacker AM, Teague J, Farrelly L, Nair A, Devaraj A, Hackshaw A, Hurst JR; SUMMIT Consortium; Janes S. Prevalence and clinical characteristics of non-malignant CT detected incidental findings in the SUMMIT lung cancer screening cohort. BMJ Open Respir Res. 2023 Jun;10(1):e001664. doi: 10.1136/bmjresp-2023-001664. PMID 37321665
- [Derived] Dickson JL, Hall H, Horst C, Tisi S, Verghese P, Mullin AM, Teague J, Farrelly L, Bowyer V, Gyertson K, Bojang F, Levermore C, Anastasiadis T, McCabe J, Navani N, Nair A, Devaraj A, Hackshaw A, Quaife SL, Janes SM; SUMMIT consortium. Uptake of invitations to a lung health check offering low-dose CT lung cancer screening among an ethnically and socioeconomically diverse population at risk of lung cancer in the UK (SUMMIT): a prospective, longitudinal cohort study. Lancet Public Health. 2023 Feb;8(2):e130-e140. doi: 10.1016/S2468-2667(22)00258-4. PMID 36709053
- [Derived] Bhamani A, Horst C, Bojang F, Quaife SL, Dickson JL, Tisi S, Hall H, Verghese P, Creamer A, Prendecki R, McCabe J, Gyertson K, Bowyer V, El-Emir E, Cotton A, Mehta S, Levermore C, Mullin AM, Teague J, Farrelly L, Nair A, Devaraj A, Hackshaw A; SUMMIT consortium; Janes SM. The SUMMIT Study: Utilising a written 'Next Steps' information booklet to prepare participants for potential lung cancer screening results and follow-up. Lung Cancer. 2023 Feb;176:75-81. doi: 10.1016/j.lungcan.2022.12.006. Epub 2022 Dec 24. PMID 36621036
- [Derived] Creamer AW, Horst C, Dickson JL, Tisi S, Hall H, Verghese P, Prendecki R, Bhamani A, McCabe J, Gyertson K, Mullin AM, Teague J, Farrelly L, Hackshaw A, Nair A; SUMMIT consortium; Devaraj A, Janes SM. Growing small solid nodules in lung cancer screening: safety and efficacy of a 200 mm3 minimum size threshold for multidisciplinary team referral. Thorax. 2023 Feb;78(2):202-206. doi: 10.1136/thorax-2022-219403. Epub 2022 Nov 25. PMID 36428100
- [Derived] Dickson JL, Bhamani A, Quaife SL, Horst C, Tisi S, Hall H, Verghese P, Creamer A, Prendecki R, McCabe J, Gyertson K, Bowyer V, El-Emir E, Cotton A, Mehta S, Bojang F, Levermore C, Mullin AM, Teague J, Farrelly L, Nair A, Devaraj A, Hackshaw A, Janes SM; SUMMIT consortium. The reporting of pulmonary nodule results by letter in a lung cancer screening setting. Lung Cancer. 2022 Jun;168:46-49. doi: 10.1016/j.lungcan.2022.04.009. Epub 2022 Apr 20. PMID 35487105